CLINICAL TRIAL: NCT05688826
Title: Comparison of Sugar Load Between Normal and Functional Variants of Sucrase-isomaltase Genes in IBS
Brief Title: The Effect of Sugar Load in IBS Patients Depending on Sucrase-isomaltase Genes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Bodil Ohlsson, Professor, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sugarload-2023
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Sucrase-Isomaltase Deficiency; Irritable Bowel Syndrome
Keywords: gastrointestinal symptoms, glucose
MeSH Terms: conditions — Sucrase-isomaltase deficiency, congenital; Irritable Bowel Syndrome | interventions — Sugars

STUDY DESIGN:
Intervention Model Description: Patients with normal genes and with functional variants of sucrase-isomaltase genes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sugar load (Experimental): Sugar dissolved in water will be ingested during 5 minutes
  Interventions: Dietary Supplement: Sugar

INTERVENTIONS:
Dietary Supplement: Sugar — 75 g sugar dissolved in 0.8 dl water and flavored with lemon. Ingested during 5 minutes

SUMMARY:
The investigators know that many patients with irritable bowel syndrome (IBS) have functional variants of genes coding for sucrase-isomaltase enzymes. The investigators will now examine whether these functional variants are associated with defect degradation of sucrose and associated gastrointestinal symptoms

DETAILED DESCRIPTION:
The investigators have in a previous study included IBS patients for treatment with a starch- and sucrose reduced diet (SSRD). The investigators found a great improvement of symptoms. The investigators gene-tested those patients, and now have the full identification of all functional variants encoding sucrase-isomaltase enzymes.

The investigators will invite patients from this previous study with normal genes and functional variants of genes. The patients will come fasting over night to the department of clinical research. The participants will ingest 75 g sugar dissolved in 0.8 dl water and flavored with lemon, to ingest during 5 minutes. After that, glucose will determined repeatedly up to 2 hours afterwards. At the same time, the participants have to assess their gastrointestinal sympotms on visual analogue scales (VAS).

The investigators will compare the raise in b-glucose and symptoms between the groups of patients, divided into gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Participants of our previous clinical trial with SSRD diet (NCT03306381)

Exclusion Criteria:

* Difficulties in taking blood samples

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of blood glucose levels | From distribution repeatedly up to 2 hours
  Measurement of glucose levels in blood drawn from an intravenous needle and analyzed at the Department of Clinical Chemostry
Change from baseline of gastrointestinal symptoms | From baseline and up to 2 hours, at the same time points as blood glucose is measured
  Measurment of gastrointestinal symptoms on a visual analog scale measuring symptoms, range 0-100 mm, repeatedly at the same time points as blood glucose is measured. The higher scores, the worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Kennback, Nurse, Study Director — Department of Internal Medicine, Skåne University Hospital, Malmö
Locations (1):
- Department of Internal Medicine, Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No